CLINICAL TRIAL: NCT03160677
Title: Comparison of Two Strategies for Blood Pressure Control in the Setting of Acute Ischemic Stroke to Reduce Cerebral Hemorrhage After Thrombectomy: Systolic Blood Pressure Target of Less Than 130 mmHg vs Less Than 185 mmHg, for 24 Hours Following Reperfusion, in Patients With Cerebral Infarction Due to Occlusion of the Anterior Circulation
Brief Title: Blood Pressure Target in Acute Stroke to Reduce hemorrhaGe After Endovascular Therapy
Acronym: BP-TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MMI_2016_26
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Acute Stroke; Blood Pressure; Cerebral Hemorrhage
Keywords: Acute Stroke; Blood Pressure; Cerebral Hemorrhage
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive blood pressure management (Experimental)
  Interventions: Other: Systolic blood pressure target < 130 mm Hg
- Standard blood pressure management (Active Comparator)
  Interventions: Other: Systolic blood pressure target < 185 mm Hg

INTERVENTIONS:
Other: Systolic blood pressure target < 130 mm Hg — Adaptation of antihypertensive treatments to reach the Systolic blood pressure target < 130 mm Hg
  Arms: Intensive blood pressure management
Other: Systolic blood pressure target < 185 mm Hg — Adaptation of antihypertensive treatments to reach the Systolic blood pressure target < 185 mm Hg
  Arms: Standard blood pressure management

SUMMARY:
A randomized, multicenter study comparing two strategies: 1 / standard management of systolic blood pressure according to international recommendations (systolic blood pressure <185 mm Hg) versus 2 / intensive blood pressure management Systolic with a target <130 mm Hg.

DETAILED DESCRIPTION:
Patients will be followed for 3 months:

* inclusion after reperfusion: clinical evaluation with NIHSS (National Institute of Health Stroke Score) score, measurement of blood pressure.
* within 24 hours after reperfusion: blood pressure measurements
* at 24 hours: measurement of blood pressure (T0 + 24 h and evaluation of the NIHSS score.
* Between 24 and 36 hours :cerebral scan (assessment of hemorrhagic transformations and cerebral infarction volumes). For some centers: Cerebral MRI without injection between H24 and H36
* 72 hours after reperfusion: Cerebral scanner in case of hyperdensity on the initial scanner
* 3 months after reperfusion: disability assessment by Rankin score

ELIGIBILITY:
Inclusion Criteria:

* Intracranial Occlusion of internal carotid arteries and/or proximal middle cerebral (segment M1) diagnosis made on initial Imaging.
* Reperfusion after a thrombectomy procedure (defined by a 2b-3 TICI score -Thrombolysis In Cerebral Infarction- score).

Exclusion Criteria:

* Per-procedure hemorrhagic complications (prior to reperfusion)
* Systolic blood pressure at baseline <130 mm Hg within one hour of recanalization
* Pre-existing stroke handicap defined by a Rankin score (modified scale, mRS)> 3
* Hemodynamically significant carotid stenosis
* Occlusion of the isolated cervical carotid artery
* Known pregnancy
* Legal protection
* Non-affiliation to a social security scheme
* Refusal of the patient (or of his / her relatives in case of urgent inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of patients with intracranial hemorrhagic complications | Scan performed between 24 and 36 hours after thrombectomy
  Rate of patients with intracranial hemorrhagic complications (Symptomatic or asymptomatic) on cerebral scan, evaluated with a double centralized blind reading

CONTACTS AND LOCATIONS:
Overall Officials: Mikael MAZIGHI, MD PhD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (7):
- France (7):
  - CHU de Bordeaux, Bordeaux
  - Hôpital neurologique Pierre Wertheimer, Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Régional Universitaire, Nancy
  - Hopital Lariboisière, Paris
  - Fondation Ophtalmologique A de Rothschild, Paris
  - Hopital Foch, Suresnes
  - Hopital de purpan, Toulouse

REFERENCES:
- [Derived] Maier B, Brauner R, Escalard S, Gory B, Lapergue B, Sibon I, Richard S, Labreuche J, Kyheng M, Desilles JP, Blanc R, Piotin M, Halimi JM, Mazighi M; BP-TARGET Trial Investigators. Association of Contrast Enhancement After Reperfusion With Outcomes According to Blood Pressure Lowering in Patients With Acute Ischemic Stroke. Neurology. 2022 Nov 22;99(21):e2385-e2394. doi: 10.1212/WNL.0000000000201173. Epub 2022 Aug 30. PMID 36041869
- [Derived] Maier B, Gory B, Lapergue B, Sibon I, Richard S, Kyheng M, Labreuche J, Desilles JP, Blanc R, Piotin M, Mazighi M, Halimi JM; BP TARGET Investigators. Effect of Baseline Antihypertensive Treatments on Stroke Severity and Outcomes in the BP TARGET Trial. Stroke. 2022 Jun;53(6):1837-1846. doi: 10.1161/STROKEAHA.121.037548. Epub 2022 Mar 24. PMID 35321558
- [Derived] Anadani M, Maier B, Escalard S, Labreuche J, de Havenon A, Sabben C, Lapergue B, Gory B, Richard S, Sibon I, Desilles JP, Blanc R, Piotin M, Mazighi M; of behalf the BP-TARGET Study Group*. Magnitude of Blood Pressure Change After Endovascular Therapy and Outcomes: Insight From the BP-TARGET Trial. Stroke. 2022 Mar;53(3):719-727. doi: 10.1161/STROKEAHA.121.036701. Epub 2022 Feb 3. PMID 35109685
- [Derived] Mazighi M, Richard S, Lapergue B, Sibon I, Gory B, Berge J, Consoli A, Labreuche J, Olivot JM, Broderick J, Duhamel A, Touze E, Qureshi AI, Yavchitz A, Escalard S, Desilles JP, Redjem H, Smajda S, Fahed R, Hebert S, Maier B, Delvoye F, Boursin P, Maacha MB, Obadia M, Sabben C, Blanc R, Savatovsky J, Piotin M; BP-TARGET investigators. Safety and efficacy of intensive blood pressure lowering after successful endovascular therapy in acute ischaemic stroke (BP-TARGET): a multicentre, open-label, randomised controlled trial. Lancet Neurol. 2021 Apr;20(4):265-274. doi: 10.1016/S1474-4422(20)30483-X. Epub 2021 Feb 26. PMID 33647246